CLINICAL TRIAL: NCT04768894
Title: Impact of Time to Re-staging Transurethral Resection on Recurrence and Progression Rates in Patient With High-risk Non-muscle-invasive Bladder Cancer: A Prospective, Randomized, Controlled Study
Brief Title: Impact of Time to Re-staging Transurethral Resection on Recurrence and Progression Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Omer Gokhan Doluoglu, Associate Professor in Urology, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SBUATRH
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Restaging transurethral resection
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a clinical study. Patients with high grade non-muscle invasive bladder canser divided three groups according to time lapse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 14-28 days (Active Comparator): In group 1,the time interval between initial and re-TUR was 14-28 days,
  Interventions: Procedure: Second transurehral resection of bladder tumour
- 29-42 days (Active Comparator): In group 2, the time interval between initial and re-TUR was 29-42 days
  Interventions: Procedure: Second transurehral resection of bladder tumour
- 43-56 days (Active Comparator): In group 3, the time interval between initial and re-TUR was 43-56 days
  Interventions: Procedure: Second transurehral resection of bladder tumour

INTERVENTIONS:
Procedure: Second transurehral resection of bladder tumour — Remove of the bladder tumour as endoscopically

SUMMARY:
Purpose To investigate the significance of time to re-staging transurethral resection (re-TUR) on recurrence and progression rates in patient with high-risk non-muscle-invasive bladder cancer.

Methods Patients diagnosed with primary high risk non-muscle-invasive bladder cancer were included to the study. The patients were randomly seperated into 3 groups acoording to Re-TUR timing. In group 1,2, and 3, the time interval between initial and re-TUR were 14-28 days, 29-42 days, and 43-56 days respectively. Kaplan -meier plots were used to estimate differences in recurrence free survival (RFS) and progression free survival (PFS) rates. Cox regression analysis was used to assess the effect of time from initial TUR to re-TUR on oncological outcomes.

Results A total of 109 patients with high risk non-muscle-invasive bladder cancer were randomly divided into 3 groups. Twenty patients in group 1 (14-28 days), 22 patients in group 2 (29-42 days), and 29 patients in group 3 (43-56 days) completed the study. The mean follow-up was 20 ± 8.9 months. Kaplan-Meier plots showed no differences in RFS and PFS rates between the three groups. Cox regression analysis demonstrated that only tumor number was found to be a prognostic factor on RFS rates.

Conclusion Our prospective study demonstrated that time laps from initial TUR to re-TUR did not significantly affect on RFS and PFS rates.

DETAILED DESCRIPTION:
This study was performed between August 2016 and December 2020 after obtaining the approval of local ethics committee (0651-5479). Patients diagnosed with primary high risk non-muscle-invasive bladder cancer at our clinic as well as the patients who were referred to our clinic with the same diagnosis were included to the study. All patients gave their written informed consent. The patients were randomly separated into 3 groups according to Re-TUR timing with the random number table envelope method. The names of the groups were written on small papers with the same size, they were folded, put in an envelope, and drawn by the doctors. In group 1,2, and 3, the time interval between initial and re-TUR were 14-28 days, 29-42 days, and 43-56 days respectively. Separate analysis was also performed for patients who had re-TUR at ≤ 42 and >42 days. All patients received six weekly instillations of BCG therapy, and at least 1 year of maintenance BCG therapy (3 weekly instillations administered at 3, 6, 12 months).

Patients with a tumor pathology other than transitional cell carcinoma, incomplete resection at initial TUR, who cannot complete 1 year of maintenance BCG treatment, did not attend their regular cystoscopic control or wanted to leave from the study voluntarily and lastly, with a diagnosis of muscle-invasive cancer on re-TUR were excluded. Inclusion criteria were having a high grade Ta or T1 transitional cell carcinoma with or without carcinoma in situ (CIS) after a complete initial TUR of bladder carcinoma, and receiving six weekly induction BCG therapy with at least 1 year maintenance.

Re-TUR contained resection of all visible tumor, deep resection of previously resected areas and adequate sampling of muscle layers. Cystoscopic control was performed according to EAU guideline recommendations for high-risk non-muscle-invasive bladder cancer [5,6]. Progresson was defined as an increase in the pathological stage (Ta to T1 or T1 to T2).

Demographic data of the patients like age, gender, and parameters related to bladder cancer such as tumor grade, T stage, concomitant CIS, number of tumors, main tumor size, application of early single dose chemotherapy, recurrence and progression were noted. Primary end points of the current study were recurrence free survival (RFS) and progression free survival (PFS) rates. Pathologic investigations were made by single expert uropathologist at our hospital.

The data analyses were performed with PASW 18 (SPSS, IBM, Chicago, IL) software. Kolmogorov-Smirnov and P-P plot tests were used to verify the normality of the distribution of continuous variables. The results were reported as means standard deviations, or in situations in which the distributions were skewed, as the median (minimum-maximum). Categorical variables were given as percentages. For parameters that did not show normal distribution, the nonparametric Kruskal Wallis One Way analysis of variance was used to compare them. Multivariable semi-parametric Cox regression analysis was used to evaluate predictors of RFS and PFS rates. Kaplan-Meier curves were constructed for RFS and PFS and groups were compared with the long-rank test. The study power and sample size were calculated with G power 3.1.9.7 version (A priori). When effect size is set to 0.33 (medium size) with 80% power, the total number of patients required to be included in the study was 73. A p value <0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a tumor pathology other than transitional cell carcinoma, incomplete resection at initial TUR, who cannot complete 1 year of maintenance BCG treatment, did not attend their regular cystoscopic control or wanted to leave from the study voluntarily and lastly, with a diagnosis of muscle-invasive cancer on re-TUR were excluded.

Exclusion Criteria:

* Inclusion criteria were having a high grade Ta or T1 transitional cell carcinoma with or without carcinoma in situ (CIS) after a complete initial TUR of bladder carcinoma, and receiving six weekly induction BCG therapy with at least 1 year maintenance.

Ages: 44 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | at least 1 year
  Recurrence free survival

IPD SHARING:
Plan to Share IPD: No